CLINICAL TRIAL: NCT04531800
Title: The Effect of Concentrated Growth Factor (CGF) in Surgical Treatment of Medication-related Osteonecrosis of the Jaw (MRONJ) in Osteoporosis Patients: a Randomized Controlled Study
Brief Title: Surgical Management of Medication Related Osteonecrosis of the Jaws With Concentrated Growth Factor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Lecturer, Ege University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: School of Dentistry
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Healing Surgical Wounds; Infection
Keywords: osteonecrosis; osteoporosis; concentrated growth factor
MeSH Terms: conditions — Infections; Osteonecrosis; Osteoporosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): The necrotic bone was removed with rotating burs, curettage was performed, and the surface of the bone was smoothened. CGF was then applied to the surgical area in the study group (n=14), and the area was primarily closed after additional releasing incisions were made to the periosteum to assure tension-free soft tissue closure.
  Interventions: Procedure: Concentrated growth factor
- Control Group (Experimental): The surgical area was only primarily closed without any mobilization of the flap following sequestrectomy and bone curettage as a traditional surgical therapy, in the control group (n=14).
  Interventions: Procedure: Non-concentrated growth factor

INTERVENTIONS:
Procedure: Concentrated growth factor — In the concentrated growth factor (CGF) group, CGF was applied to the surgical area (n=14), and the area was primarily closed after additional releasing incisions.
  Arms: Study Group
Procedure: Non-concentrated growth factor — In the non-CGF group, the surgical area was only primarily closed without any mobilization of the flap following sequestrectomy and bone curettage as a traditional surgical therapy.
  Arms: Control Group

SUMMARY:
The purpose of this present study was to evaluate the efficiency of the growth factors delivered by concentrated growth factor (CGF) on the healing process of osteoporotic patients with medication-related osteonecrosis of the jaws (MRONJ).

This randomized controlled study composed of osteoporotic female patients who were treated with oral bisphosphonates (BPs) and diagnosed with MRONJ. For the CGF group, each patient was treated with local application of CGF at the surgical site after removing the necrotic bone while the surgical area was only primarily closed as traditional surgical therapy for the control group. The patients underwent clinical examinations for 6 months postoperatively to check the presence of infection and dehiscence.

DETAILED DESCRIPTION:
This randomized controlled study comprised 28 elderly female osteoporotic patients diagnosed with MRONJ at the department of oral and maxillofacial surgery of a university hospital between May 2016 and April 2018.

Before the surgery, the sequentially numbered sealed envelopes were used to randomly assign patients to the study groups:

Study group (14 patients treated with CGF clots + primarily closure) Control group (14 patients treated without CGF placement + primarily closure)

All procedures were performed under local anesthesia by the same surgeon. After removal of superficial bone sequestrum, the necrotic bone was removed with rotating burs, curettage was performed, and the surface of the bone was smoothened (Fig. 2). CGF was then applied to the surgical area in the study group (n=14), and the area was primarily closed after additional releasing incisions were made to the periosteum to assure tension-free soft tissue closure (Fig. 3). In the control group (n=14), the surgical area was only primarily closed without any mobilization of the flap following sequestrectomy and bone curettage as a traditional surgical therapy. A soft diet and daily irrigation with 0.12% chlorhexidine were prescribed for 2 weeks postoperatively. The sutures were removed 14 days postoperatively.

The primary outcome variable of this study was soft tissue healing 6 months post-operatively. The patients underwent weekly clinical examinations for the 1st month and then monthly clinical examinations for 6 months postoperatively. At the time of the evaluation, soft tissue coverage in the surgical site was assessed without signs of infection and/or necrotic bone. The presence of infection was assessed as follows: erythema, swelling, bleeding on probing and purulent exudate. The differences between the study groups were recorded and considered to indicate postoperative healing. BP treatment status and ONJ classification of each patient were recorded and these differences were also assessed in soft tissue healing.

In addition, anamnestic and therapeutic data as patients' age, the type of BPs, timing of medication, location of the exposed necrotic bone and MRONJ-promoting factors were recorded for each patient.

ELIGIBILITY:
Inclusion Criteria:

1. treatment with oral bisphosphonates (BPs) for osteoporosis,
2. MRONJ diagnosis with exposed bone in the jaws that had persisted for longer than 8 weeks according to 2014 recommendations of the Association of Oral and Maxillofacial Surgeons (AAOMS),
3. MRONJ stage 2 or 3 with bone destruction and sequestrum confirmed by clinical and radiographic examination,
4. insufficient improvement with conservative treatment.

Exclusion Criteria:

1. a history of head and neck radiation therapy,
2. metastatic bone disease of the jaws,
3. platelet values under than 150,000 mm3 in a complete blood count.

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Because of the large number of cases of osteoporosis and breast cancer, MRONJ was found to be more common in women.
Enrollment: 28 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Soft tissue healing | Change of soft tissue healing 6 months postoperatively
  Healing was defined as the previous studies. The patients underwent weekly clinical examinations for the 1st month and then monthly clinical examinations for 6 months postoperatively. At the time of the evaluation, soft tissue coverage in the surgical site was assessed without signs of infection and/or necrotic bone. The presence of infection was assessed as follows: erythema, swelling, bleeding on probing and purulent exudate.

CONTACTS AND LOCATIONS:
Overall Officials: Gözde Işık, Principal Investigator — Lecturer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beth-Tasdogan NH, Mayer B, Hussein H, Zolk O, Peter JU. Interventions for managing medication-related osteonecrosis of the jaw. Cochrane Database Syst Rev. 2022 Jul 12;7(7):CD012432. doi: 10.1002/14651858.CD012432.pub3. PMID 35866376